CLINICAL TRIAL: NCT00510861
Title: Influence of Paternal Age on Assisted Reproduction Outcome
Acronym: MALE AGING
Status: Completed | Type: Observational
Sponsor: Instituto Valenciano de Infertilidad, IVI VALENCIA (Other)
Other Study IDs: VLC-MM-0205-507-26
Record Dates: First submitted 2007-08-01; First posted 2007-08-02 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: We Will Retrospectively Assess Our Databases in Our Clinic; Instituto Valenciano de Infertilidad in Valencia (Spain); Searching for Assisted Reproduction Procedures; IUI Standard IVF/ICSI Cycles and Ovum Donation IVF/ICSI Cycles; Who Were Referred to Our Unit to Cryopreserve Sperm During the Period; From January 2000 to December 2006
Keywords: male age, assisted reproduction, sperm, pregnancy outcome

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
In the recent years, there is an increasing tendency to the parenthood delay in developed countries, and there is not enough information available regarding the influence of the male's age on fertility. If any, the negative impact should be acting at advanced ages.

Our aim with this work was to determine the role of paternal age on IUI results embryo quality and IVF outcome. Evenmore, in order to standardize the female factor, good quality oocytes (from fertile oocyte donors) and only first IVF cycles in young women were considered.

DETAILED DESCRIPTION:
A retrospective study has been designed with a total number of 2204 IUI, 1286 IVF cycles and 1412 IVF cycles with donated oocytes from 2000 to 2006.

The inclusion criteria will be for IUI: women under 38 years old, tubal patency demonstrated by hysterosalpingography, normal uterine scan, normal basal hormonal levels, body mass index < 27 kg/m2, and absence of polycystic ovarian syndrome and endometriosis. For normal IVF cycles and oocyte donation cycles only first cycles will be analyzed. Cycles will be studied only in couples with absence of severe male factor.

ELIGIBILITY:
Inclusion Criteria:

* women under 38 years old, tubal patency demonstrated by hysterosalpingography, normal uterine scan, normal basal hormonal levels, body mass index < 27 kg/m2.

Exclusion Criteria:

* absence of polycystic ovarian syndrome, hydrosalpinx or endometriosis.
* Cycles were studied only in couples with absence of severe male factor.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2007-02; Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marcos Meseguer, PhD, Principal Investigator — IVI Valencia
Locations (1):
- IVI, Valencia, Spain